CLINICAL TRIAL: NCT07250295
Title: The Effect of Exercise on Paravertebral Muscle Thickness and Quality of Life in Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Roza Jizel Dagdelen MD, MD, Principal Investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 28.12.2021 / 3388
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Exercise; Muscles; Scoliosis; Ultrasound
MeSH Terms: conditions — Motor Activity; Scoliosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): The treatment group (TG) was given exercises for the thoracic and lumbar regions for scoliosis.
  Interventions: Other: Exercise
- Control Group (Placebo Comparator): The control group (CG) was instructed to perform gluteus maximus, hamstring, and quadriceps strengthening exercises.
  Interventions: Other: Exercise for Lower Extremities

INTERVENTIONS:
Other: Exercise — Patients were expected to attend treatment under the supervision of a physiotherapist. If they missed a day, they were contacted by phone and advised to do their exercises at home. The number of days they missed did not exceed five. Each set included a 30-second rest period to prevent fatigue. A five-minute warm-up and cool-down period was allotted before and after the exercise session. The exercise program was implemented by a physiotherapist with three years of experience in scoliosis management. Before initiating the intervention, the physiotherapist underwent a structured training session, including practical demonstrations, supervised practice, and detailed exercise protocols.
  Arms: Treatment Group
Other: Exercise for Lower Extremities — The control group (CG) was instructed to perform gluteus maximus, hamstring, and quadriceps strengthening exercises.
  Arms: Control Group

SUMMARY:
The study population comprised patients with AIS who had applied to the outpatient clinic between January and June 2022. The patients were divided into two groups. Treatment group(TG) was instructed in specific scoliosis exercises, while the Control group(CG) was given exercises for the lower extremities. Each patient was included in a 12- week exercise program accompanied by a physiotherapist. The patients' quality of life, and paravertebral muscles were evaluated ultrasonographically before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had been diagnosed with AIS by means of radiographic and clinical examination of the spine were included in the study.

Exclusion Criteria:

* Cases with a history of surgery to the paravertebral region
* Metabolic bone disease
* Neuromuscular disease
* chromosomal anomaly
* Serious autoimmune and endocrine disease
* Congenital scoliosis
* Skeletal dysplasia and serious cognitive impairment

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Paravertebral Muscle Thickness in Ultrasonographic Measurements | 12 weeks
  A standard imaging protocol was employed for the transverse imaging of the thoracic and lumbar multifidus muscles. Pre- and post-exercise measurements were performed by the same physician who was blinded to the exercise program the patient received. This evaluator was a PMR physician with 3 years of experience in the field of ultrasound. For each ultrasound image, the examiner positioned the probe over the spinous process and then moved it laterally and proceeded to image the multifidus and deep thoracic paravertebral muscles on both the convex and concave sides of the apex with the patient positioned prone. Two images were obtained for each segment on each side. The mean of the two trials was employed for the purpose of data analysis.
The Turkish version of the Spinal Appearance Questionnaire (Tr-SGA) | 12 weeks
  The questionnaire comprises two distinct sections: one pertaining to appearance and the other to expectations. Each section contains a series of questions presented on a 5-point Likert scale.

SECONDARY OUTCOMES:
The Short Form-36 Health Status Questionnaire (SF-36) | 12 weeks
  The Short Form-36 Health Status Questionnaire (SF-36) was employed for the purpose of assessing quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)